CLINICAL TRIAL: NCT00920075
Title: Phase II Study of Alendronate Sodium in Juvenile Osteoporosis (IND# 60,017)-Post Study Evaluation of Participants From Phase IIa and Phase IIb Clinical Study.
Brief Title: Alendronate in Juvenile Osteoporosis
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Deborah A Bowlby, MD, Assistant Professor, Medical University of South Carolina
Other Study IDs: 5R01FD001847-05 REVISED; FD-R-001847-03 (Other: FDA); 5R01FD001847-05 (NIH)
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Results first posted 2010-12-10 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2010-11

CONDITIONS: Juvenile Osteoporosis; Low Bone Density; Fractures
Keywords: Juvenile Osteoporosis; Bone Mineral Density; Fosamax; Dual Energy X-Ray Absorptiometry; Fracture
MeSH Terms: conditions — Juvenile osteoporosis; Bone Diseases, Metabolic; Fractures, Bone | interventions — Alendronate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1 Alendronate for 12 months, post study: Participants earlier were treated with alendronate for 12 months either in an open label study (without control) or double blind study with placebo control. These studies were completed. In this post study evaluation, available participants will be scheduled for one clinic visit to assess their current status of the bone density and no treatment is involved.
  Interventions: Drug: Alendronate (Fosamax)

INTERVENTIONS:
Drug: Alendronate (Fosamax) — Pill, 35mg or 70mg depending upon the body weight for 12 months. This was given for participants during the open label or double blind study. Current study is a post study evaluation of the current status of bone density after the participants completed the study. In this post study, no treatment is involved.
  Other Names: Fosamax

SUMMARY:
The investigators earlier have shown that treatment of patients with juvenile osteoporosis with alendronate (Fosamax) for 12 months increased the bone density without side effects. In an open label study (10 patients) and double blind, crossover study (11 patients alendronate and 11 patients placebo), the investigators have further observed that alendronate increased the bone density significantly where as placebo (calcium and vitamin D) increased only minimally. These trials were completed. Thus, a post study is designed to evaluate the current status of the bone density and fractures after the patients discontinued the alendronate treatment. No treatment is involved.

DETAILED DESCRIPTION:
With the availability of Dual Energy X-ray Absorptiometry (DXA), juvenile osteoporosis has been recognized and diagnosed in recent years. The disease results from either diminished bone formation or increased bone removal (resorption) resulting in low bone density and fractures. No specific drug therapy has been recommended for juvenile osteoporosis. In an open label study, we earlier have shown that alendronate treatment (10 patients) for 12 months increased bone density without side effects. Subsequently, in a double blind, crossover study, we have further confirmed that alendronate treatment (11 patients) increased bone density significantly whereas, placebo (11 patients with calcium and vitamin D), increased the bone density only minimally. There were no side effects. These patients were treated with alendronate only for 12 months and the clinical trials have been completed. We therefore, have designed a post study to evaluate the current status of the bone density and fracture history in the above participants after the discontinuation (1-6 years) of alendronate treatment. Available participants, who have completed the earlier study, will be scheduled for a one time clinic visit. Measurements include DXA bone density measurement of spine and hip, urinalysis and blood work. No treatment is involved.

ELIGIBILITY:
Inclusion Criteria:

* Participated in our earlier clinical study;
* Completed the earlier open label or double blind study;
* Availability to participate in the post study;
* Male and female children who have earlier participated in our clinical trial; AND
* Parental consent (and patient assent after age 12 years) to participate in the study. Participant's consent for those who have completed 18 years of age and above at the time of clinic visit.

Exclusion Criteria:

* Not participated in our earlier clinical study;
* Not completed our earlier trials; OR
* Pregnancy.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Available male and female children who have participated and Completed in our earlier open label or double blind clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Bowlby, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Key LL Jr, Ries W, Madyastha P, Reed F. Juvenile osteoporosis: recognizing the risk. J Pediatr Endocrinol Metab. 2003 May;16 Suppl 3:683-6. PMID 12795371
- See also: Juvenile Osteoporosis Clinical Trial — http://www.musckids.com/research/fosamax_trial.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who have completed our earlier phase-1 and II study on alendronate in juvenile osteoporosis will be invited in this post study to evaluate the bone density/ fractures after discontinuation of therapy. Interested participants will be scheduled for a one time clinic visit. No treatment is involved.
Pre-assignment Details: Participants should have completed our earlier phase I or II study on alendronate in juvenile osteoporosis. Participants will be recruited by invitation only.
Period: Last Study, 25 Pts Invited,11 Responded
Arm/Group | 1 Alendronate for 12 Months, Post Study
Started | 11
Completed | 11
Not Completed | 0
Period: Post Study, 11 Pts Responded
Arm/Group | 1 Alendronate for 12 Months, Post Study
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 1 Alendronate for 12 Months, Post Study
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.9 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density (BMD) of the Lumbar Spine (Participants With Percentage Increase).
Description: Participants who earlier completed in our open labeled or double blind study of alendronate treatment for juvenile osteoporosis, were invited for one clinical visit. Bone density of spine was measured by DXA scan.
Time Frame: Post study (1-6 yrs), one clinical visit
Population: Participants who earlier completed our phase I or phase II study on alendronate in juvenile osteoporosis, were invited to participate in the current post study evaluation of bone density and fractures.
Measure: Number; unit: participants
Arm/Group | 1 Alendronate for 12 Months, Post Study
Number analyzed (Participants) | 11
participants | 11

2. Secondary Outcome: Bone Mineral Density (BMD) of the Hip (Participants With Percentage Increase).
Description: Participants who earlier completed in our open labeled or double blind study of alendronate treatment for juvenile osteoporosis, were invited for one clinical visit. Bone density of hip was measured by DXA scan.
Time Frame: Post study (1-6 years), one clincial visit
Population: 11 participants responded to participate in the post study. Their bone density of Hip was measured by DXA scan. Increase in percentage density of Hip was obtained from that of previous values. One participant showed a slight decrease in bone density.
Measure: Number; unit: participants
Arm/Group | 1 Alendronate for 12 Months, Post Study
Number analyzed (Participants) | 11
participants | 10

3. Secondary Outcome: Number of Participants With Fracture
Description: Participants who earlier completed in our open labeled or double blind study of alendronate treatment for juvenile osteoporosis, were invited for one clinical visit. Their bone densities of spine and hip were measured by DXA scan. During this visit, their fracture history was obtained.
Time Frame: Post study (1-6 years), one clinical visit
Population: 11 participants responded to participate in the post study. During their one clinic visit, their fracture history during the period before coming to the post study was obtained.
Measure: Number; unit: participants
Arm/Group | 1 Alendronate for 12 Months, Post Study
Number analyzed (Participants) | 11
participants | 0

ADVERSE EVENTS:
Time Frame: 1-6 years post study
Description: Participants who completed our earlier phase I/II study on alendronate in juvenile osteoporosis were invited to participate in the current post study evaluation of their current bone density/fracure history. Durine their one time clinic visit, they were asked regarding any adverse events they had during the period before coming to the post study.
Arm/Group | 1 Alendronate for 12 Months, Post Study
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement with Merck: to submit a copy of any proposed abstract, manuscript and/or press release to Merck for review and comment at least 30 days prior to submission for publication or presentation.